CLINICAL TRIAL: NCT06325423
Title: The Impact of Tumor Microenvironment and Clinicopathological Features in Predicting Response to Neoadjuvant Chemotherapy in Muscle Invasive Bladder Cancer
Brief Title: Predicting Response to Neoadjuvant Chemotherapy in Muscle-invasive Bladder Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Ahmed Abd El-Razik, Assistant Lecturer, Assiut University
Other Study IDs: response to NAC in MIBC
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: MIBC
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — baseline formalin-fixed paraffin-embedded (FFPE) transurethral resection (TUR) biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MIBC patients who received NAC: Patients with muscle-invasive bladder cancer who received neoadjuvant chemotherapy before radical cystectomy or bladder preservation
  Interventions: Combination Product: neoadjuvant chemotherapy

INTERVENTIONS:
Combination Product: neoadjuvant chemotherapy — platinum-based chemotherapy before radical cystectomy or bladder preservation

SUMMARY:
Bladder cancer (BC) is the 10th most commonly diagnosed cancer worldwide and the second most common cancer among Egyptian males.

The mainstay of treatment of muscle-invasive BC( MIBC) is neoadjuvant chemotherapy (NAC) followed by radical cystectomy (RC) or bladder preservation(BP) using maximal transurethral resection of the bladder tumor followed by chemoradiation. The rationale to use NAC before RC or BP is to eradicate micro-metastasis and to downstage the primary tumor.

The 5-year cancer-specific survival for responders to NAC is 90%, in contrast to 30-40% for those not obtaining an objective response. Drawbacks of NAC are disappointing delay of surgery in non-responders and the potential toxicity. So, predictors of response to NAC are necessary to identify patients who may achieve pathologic complete response and will benefit from BP, and the others who may not respond to NAC and spare them NAC toxicity and RC delay.

Tumor microenvironment (TME), including neutrophil extracellular traps (NETs), and CD8+ T lymphocytes is a promising predictor of response to NAC in MIBC.

NETs are reticulated DNA structures decorated with various protein substances (e.g., histones, myeloperoxidase, neutrophil elastase).NETs are involved in tumor growth, metastasis, and treatment resistance. Moreover, NETs can inhibit T cell responses, thereby promoting tumor growth.

On the other hand, immune cells that are present in the TME play a major role in slowing down tumor progression. CD8+T lymphocytes play a central role in immune-mediated control of cancer . Also, they have been found to be a prognostic tool for advanced BC.

DETAILED DESCRIPTION:
Formalin fixed paraffin embedded tissue specimen of the baseline TUR of MIBC will be obtained from pathology laboratory, Pathology Department, Assiut University.

* Histological diagnosis of H&E stained sections will be confirmed.
* Immunohistochemical staining for Citrullinated histone H3 (H3Cit) antibody as a hallmark of NETs, and CD8 antibody to quantity density of NETs and CD8 expression, then calculate NETs/CD8 ratio.
* Baseline clinicopathological features of MIBC patients who received neoadjuvant chemotherapy will be collected from patients' records.
* Correlation between NETs expression, CD8 expression, NETs/CD8 ratio, and the baseline clinicopathological features with the response to neoadjuvant chemotherapy.
* develop a risk score based on the significant predictors of response to identify patients who may achieve pathologic complete response and will benefit from BP, and the others who may not respond to NAC and spare them NAC toxicity and RC delay.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven pure urothelial carcinoma, or morphologic variant of urothelial carcinoma.
* Patients with ≥T2, N0-1, M0, according to American Joint Committee on Cancer (AJCC) TNM Staging System for Bladder Cancer 8th ed., 2017.
* Patients who received platinum-based neoadjuvant chemotherapy before RC or BP.
* Available paraffin-embedded TUR specimens for Immunohistochemistry (IHC).

Exclusion Criteria:

* Non urothelial carcinoma.
* Not muscle invasive < T2.
* Metastatic bladder cancer.
* No available paraffin-embedded TUR specimens for IHC.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with localised muscle-invasive bladder cancer who received neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the expression of NETs and CD8 in paraffin-embedded TUR biopsies | 6 months
  evaluation of the density of Citrullinated Histone H3 as a hallmark of NETs and the density of CD8 in the baseline FFPE TUR specimens
- Response to platinum-based chemotherapy in localized MIBC in relation to: NETs expression, CD8 expression, NET/CD8 ratio and baseline clinicopathological features | 6 months
  Correlation between NETs expression, CD8 expression, NETs/CD8 ratio and the baseline clinicopathological features of MIBC and the response to neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Local recurrence-free survival (RFS) | 2 years
  the length of time from radical cystectomy/ bladder preservation to local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Amal R Ibrahim, Ass.Prof, Study Director — Assiut University; Hanan G Mostafa, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Skinner DG, Lieskovsky G. Contemporary cystectomy with pelvic node dissection compared to preoperative radiation therapy plus cystectomy in management of invasive bladder cancer. J Urol. 1984 Jun;131(6):1069-72. doi: 10.1016/s0022-5347(17)50809-5. PMID 6726903
- [Result] Rosenblatt R, Sherif A, Rintala E, Wahlqvist R, Ullen A, Nilsson S, Malmstrom PU; Nordic Urothelial Cancer Group. Pathologic downstaging is a surrogate marker for efficacy and increased survival following neoadjuvant chemotherapy and radical cystectomy for muscle-invasive urothelial bladder cancer. Eur Urol. 2012 Jun;61(6):1229-38. doi: 10.1016/j.eururo.2011.12.010. Epub 2011 Dec 13. PMID 22189383
- [Result] Jiang DM, Jiang H, Chung PWM, Zlotta AR, Fleshner NE, Bristow RG, Berlin A, Kulkarni GS, Alimohamed NS, Lo G, Sridhar SS. Neoadjuvant Chemotherapy Before Bladder-Sparing Chemoradiotherapy in Patients With Nonmetastatic Muscle-Invasive Bladder Cancer. Clin Genitourin Cancer. 2019 Feb;17(1):38-45. doi: 10.1016/j.clgc.2018.09.021. Epub 2018 Oct 4. PMID 30686350
- [Result] Witjes JA, Comperat E, Cowan NC, De Santis M, Gakis G, Lebret T, Ribal MJ, Van der Heijden AG, Sherif A; European Association of Urology. EAU guidelines on muscle-invasive and metastatic bladder cancer: summary of the 2013 guidelines. Eur Urol. 2014 Apr;65(4):778-92. doi: 10.1016/j.eururo.2013.11.046. Epub 2013 Dec 12. PMID 24373477
- [Result] Ikarashi D, Kitano S, Tsuyukubo T, Takenouchi K, Nakayama T, Onagi H, Sakaguchi A, Yamashita M, Mizugaki H, Maekawa S, Kato R, Kato Y, Sugai T, Nakatsura T, Obara W. Pretreatment tumour immune microenvironment predicts clinical response and prognosis of muscle-invasive bladder cancer in the neoadjuvant chemotherapy setting. Br J Cancer. 2022 Mar;126(4):606-614. doi: 10.1038/s41416-021-01628-y. Epub 2021 Nov 15. PMID 34782748
- [Result] Zhao J, Jin J. Neutrophil extracellular traps: New players in cancer research. Front Immunol. 2022 Aug 19;13:937565. doi: 10.3389/fimmu.2022.937565. eCollection 2022. PMID 36059520
- [Result] Kaltenmeier C, Yazdani HO, Morder K, Geller DA, Simmons RL, Tohme S. Neutrophil Extracellular Traps Promote T Cell Exhaustion in the Tumor Microenvironment. Front Immunol. 2021 Nov 24;12:785222. doi: 10.3389/fimmu.2021.785222. eCollection 2021. PMID 34899751
- [Result] Koebel CM, Vermi W, Swann JB, Zerafa N, Rodig SJ, Old LJ, Smyth MJ, Schreiber RD. Adaptive immunity maintains occult cancer in an equilibrium state. Nature. 2007 Dec 6;450(7171):903-7. doi: 10.1038/nature06309. Epub 2007 Nov 18. PMID 18026089
- [Result] Durgeau A, Virk Y, Corgnac S, Mami-Chouaib F. Recent Advances in Targeting CD8 T-Cell Immunity for More Effective Cancer Immunotherapy. Front Immunol. 2018 Jan 22;9:14. doi: 10.3389/fimmu.2018.00014. eCollection 2018. PMID 29403496
- [Result] Hadrup S, Donia M, Thor Straten P. Effector CD4 and CD8 T cells and their role in the tumor microenvironment. Cancer Microenviron. 2013 Aug;6(2):123-33. doi: 10.1007/s12307-012-0127-6. Epub 2012 Dec 16. PMID 23242673
- [Result] Sharma P, Retz M, Siefker-Radtke A, Baron A, Necchi A, Bedke J, Plimack ER, Vaena D, Grimm MO, Bracarda S, Arranz JA, Pal S, Ohyama C, Saci A, Qu X, Lambert A, Krishnan S, Azrilevich A, Galsky MD. Nivolumab in metastatic urothelial carcinoma after platinum therapy (CheckMate 275): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2017 Mar;18(3):312-322. doi: 10.1016/S1470-2045(17)30065-7. Epub 2017 Jan 26. PMID 28131785